CLINICAL TRIAL: NCT00087204
Title: A Phase I Study Of XL119 In Patients With Relapsed Or Refractory Acute Myeloid Leukemia, Myelodysplastic Syndromes, Acute Lymphocytic Leukemia, Or Chronic Myeloid Leukemia In Blastic-Phase
Brief Title: Rebeccamycin Analog in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia, Myelodysplastic Syndrome, Acute Lymphoblastic Leukemia, or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02609; MDA-2003-0909; U01CA062461 (NIH); CDR0000373813 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — becatecarin

ARMS (1):
- Treatment (becatecarin) (Experimental): Patients receive rebeccamycin analogue (XL119) IV over 1 hour on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a CR receive 1 additional course beyond CR. Patients achieving a PR or HI receive 2 additional courses beyond PR or HI. Cohorts of 3-6 patients receive escalating doses of XL119 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: becatecarin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: becatecarin — Given IV
  Other Names: BMS-181176; rebeccamycin analogue; rebeccamycin analogue, tartrate salt; XL119
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of rebeccamycin analog in treating patients with relapsed or refractory acute myeloid leukemia, myelodysplastic syndrome, acute lymphoblastic leukemia, or chronic myelogenous leukemia in blast phase. Drugs used in chemotherapy, such as rebeccamycin analog, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicity of rebeccamycin analogue (XL119) in patients with relapsed or refractory acute myeloid leukemia, myelodysplastic syndromes, acute lymphoblastic leukemia, or chronic myelogenous leukemia in blastic phase.

OUTLINE: This is a dose-escalation study.

Patients receive rebeccamycin analogue (XL119) IV over 1 hour on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 1 additional course beyond CR. Patients achieving a partial response (PR) or hematologic improvement (HI) receive 2 additional courses beyond PR or HI. Cohorts of 3-6 patients receive escalating doses of XL119 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia
  * Myelodysplastic syndromes, including 1 of the following:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia in transformation with ≥ 10% peripheral blood or bone marrow blasts
  * Acute lymphoblastic leukemia
  * Chronic myelogenous leukemia in blastic phase
* Relapsed or refractory disease, defined as 1 of the following:

  * Failed to achieve a complete response (CR) to a standard induction regimen
  * Relapsed after achieving a CR
* Failed last cytotoxic regimen before study entry
* No alternate, potentially curative option available
* No known CNS disease
* Performance status - ECOG 0-2
* SGOT and SGPT normal
* Bilirubin normal
* Creatinine normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV-positive patients with normal CD4 count and without AIDS-defining disease allowed
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to rebeccamycin analogue (XL119)
* No concurrent uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior allogeneic stem cell transplantation
* No concurrent prophylactic hematopoietic colony-stimulating factors (CSF)
* No epoetin alfa or hematopoietic CSF during course 1 of study therapy
* More than 7 days since prior cytotoxic chemotherapy except for hydroxyurea
* More than 7 days since prior radiotherapy
* Recovered from all prior therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No other concurrent antileukemic agents or therapies
* No other concurrent investigational agents or therapies
* No other concurrent cytotoxic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of becatecarin | 21 days
  Graded using the NCI CTCAE version 3.0.

SECONDARY OUTCOMES:
Survival | From date of first study drug administration to the date of death of the patients, assessed up to 3 years
Time to progression | From the date of first study drug administration to the date that the patient is withdrawn because of clinical or radiographic progressive disease, or death from any cause, assessed up to 3 years
Time to treatment failure | From the date of first study drug administration to the date of withdrawal from the study for any reason other than study closure, assessed up to 3 years
Duration of response | From the date of first objective response to the date of progression, assessed up to 3 years
Time to response | From the date of first study drug administration until the first objective documentation of response, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis Giles, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States